CLINICAL TRIAL: NCT03002649
Title: Study of Tofacitinib in Refractory Dermatomyositis (STIR): Proof of Concept, Open-Label Study of 10 Patients
Brief Title: Study of Tofacitinib in Refractory Dermatomyositis
Acronym: STIR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00084227
Record Dates: First submitted 2016-12-20; First posted 2016-12-26 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-06

CONDITIONS: Dermatomyositis
Keywords: Dermatomyositis; Tofacitinib; Refractory dermatomyositis
MeSH Terms: conditions — Dermatomyositis | interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tofacitinib (Experimental): All subjects will be provided Tofacitinib 11mg tablets for oral administration once daily. 12-week treatment period with optional 4-week treatment extension period.
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Tofacitinib — Tofacitinib comes as an extended-release (XR) (long-acting) tablet to take by mouth. The extended-release tablet is usually taken with or without food once daily.
  Other Names: Xeljanz XR; Tofacitinib citrate

SUMMARY:
The purpose of this study is to obtain preliminary data regarding the safety and efficacy of Janus kinase (JAK) inhibitor, tofacitinib, in adults with active, treatment-refractory dermatomyositis.

DETAILED DESCRIPTION:
Dermatomyositis (DM) is a rare, progressively debilitating disorder that affects the muscle (causing weakness) and skin (causing a rash) in most affected patients. DM can also involve multiple body systems including the lungs, joints, gut and heart. Therapy for DM involves administering corticosteroids, typically with an immunosuppressive agent, but treatment options for refractory DM are very limited. This research is being done to determine the safety and effectiveness of a Janus kinase (JAK) inhibitor called Tofacitinib in adults with active, treatment-refractory dermatomyositis. The investigators will also look for specific biomolecular changes in blood, skin, and muscle when it is exposed to Tofacitinib. Tofacitinib is approved by the Food and Drug Administration (FDA) for the treatment of rheumatoid arthritis. The study aim is to conduct a 12-week, open-label, pilot study with up to 10 patients who have refractory DM to assess whether a JAK inhibitor effectively and safely reduces the symptoms of DM in both the skin and muscle. This study consists of up to 9 study visits over 6 months. There is an optional treatment extension period of 4 weeks. All subjects will undergo follow-up assessments 4 weeks after stopping treatment. Results from this study will contribute to the design of future trials that will further define the role of JAK inhibitors in the treatment of patients with dermatomyositis.

ELIGIBILITY:
Inclusion Criteria:

Study subjects must meet the following criteria:

* Definite or probable dermatomyositis by Bohan and Peter Criteria at least 6 months before screening
* Active skin disease as defined by a CDASI score of at least 5
* Skin biopsy proven disease
* Although not mandatory, patients with muscle weakness are eligible for enrollment. Those with active muscle disease must have a Manual Muscle Testing (MMT-8) score < 142 out of 150
* Age > 18
* Refractory myositis is defined by active disease despite a 12 week trial of steroids and with failure of response to at least prednisone and 1 other first line immunosuppressive agents (e.g. methotrexate, mycophenolate mofetil, or azathioprine) OR have demonstrated significant toxicity or intolerance to such therapies
* Maximum prednisone dose allowed will be 20mg/daily at time of entry to study provided that the dose has been stable for at least 2 weeks prior to baseline. Patients should not have received a daily therapy of more than 80mg of prednisone equivalent within 8 weeks prior to study entry
* Negative cancer screening conducted in the 6 months prior to screening visit
* Washout of immunosuppressive agents will be as follows:

  1. Azathioprine, mycophenolate, tacrolimus: 12-16 weeks prior to first dose of study drug;
  2. Rituximab: 12 months;
  3. Intravenous Immunoglobulin (IVIg): 3 months;
  4. Cyclophosphamide: 1 year;
  5. Methotrexate: 12-16 weeks.
* Women of child-bearing potential must have negative pregnancy test and be willing to undergo urine pregnancy testing at every on-site visit for the duration of the study
* Must provide informed consent
* Must be willing and able to comply with the requirements of the protocol

Exclusion Criteria:

The presence of any of the following excludes subject participation in the study:

* Use of other investigational drugs at the time of enrollment
* History of hypersensitivity to any of the study drugs or drugs of similar chemical classes
* DM patients having overlap myositis attributable to other causes such as scleroderma, arthritis, statin myopathy, steroid induced myopathy and/or significant organ damage e.g. lupus nephritis, central nervous system are present
* Late stage DM whose muscle weakness, according to the Investigator, could be attributable to muscle damage rather than myositis disease activity
* Patients with other types of myositis or myopathies: polymyositis, paraneoplastic myositis, inclusion body myositis, metabolic or drug induced myopathy, dystrophies
* Inclusion body myositis, Juvenile dermatomyositis or polymyositis, or myositis in overlap with other rheumatic diseases such as lupus, scleroderma, Sjogren's, or vasculitis
* Patients with advanced clinically symptomatic interstitial lung disease
* Pregnancy or breast-feeding patients
* History of bowel rupture or inflammatory bowel diseases
* History of tuberculosis or mycobacterial infections
* Recent infection in the past 4 weeks before entry of study
* History of any malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases
* Active systemic bacterial, viral or fungal infections, or diagnosis of AIDS, Hepatitis B, Hepatitis C infection
* Diverticulitis or ulcers in stomach or intestines
* Evidence of any other acute or chronic infectious diseases
* Have received any live or live attenuated vaccines (including varicella or measles) within 2 months prior to study enrollment
* Patients with any of the following hepatic conditions prior to study: (a) history of chronic liver or biliary disease, (b) total conjugated bilirubin greater than 1.5 times upper limits of normal (ULN) range, unless in the context of Gilbert's syndrome, (c) alkaline phosphatase greater than 1.5 times the ULN range, (d) aspartate transaminase (AST), alanine transaminase (ALT) greater than 3 times the ULN if the elevation of AST or ALT, according to the investigator, is attributable to liver disease. Patients with elevated AST/ALT due to myositis disease activity are eligible, (e) Gamma-glutamyltransferase (GGT) greater than 3 times the ULN range
* Current or recent history of uncontrolled renal, hepatic, hematological, gastrointestinal, metabolic, endocrine, pulmonary, cardiac, or neurological disease
* Blood dyscrasias within 3 months prior to the first dose of study medication, including confirmed:

  1. Hemoglobin <9 g/dL or Hematocrit <30%;
  2. White blood cell count <3.0 x 109/L;
  3. Absolute neutrophil count <1.2 x 109/L;
  4. Platelet count <100 x 109/L.
* Estimated glomerular filtration rate (GFR) <40 ml/min based on Cockcroft-Gault calculation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-01; Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Number of participants who achieve International Myositis Assessment and Clinical Studies (IMACS) Definition of Improvement (DOI) | Up to 12 weeks
  IMACS DOI is 3 of any of the 6 core set measures (CSM) improved by ≥ 20%, with no more than 2 CSM worsening by ≥25% (worsening measure cannot include the manual muscle testing)

SECONDARY OUTCOMES:
Change from baseline in CDASI activity score | Up to 16 weeks
Safety and tolerability of tofacitinib as assessed by frequency of adverse events reported and observed | Up to 16 weeks
Safety and tolerability of tofacitinib as assessed by incidence of adverse events reported and observed | Up to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Julie Paik, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paik JJ, Casciola-Rosen L, Shin JY, Albayda J, Tiniakou E, Leung DG, Gutierrez-Alamillo L, Perin J, Florea L, Antonescu C, Leung SG, Purwin G, Koenig A, Christopher-Stine L. Study of Tofacitinib in Refractory Dermatomyositis: An Open-Label Pilot Study of Ten Patients. Arthritis Rheumatol. 2021 May;73(5):858-865. doi: 10.1002/art.41602. Epub 2021 Mar 24. PMID 33258553